CLINICAL TRIAL: NCT02952079
Title: Comparison of BlephEx to MiBoflo as Treatment Options for Blepharitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Principal Investigator, SRIHARI NARAYANAN, Professor, University of the Incarnate Word
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-06-015
Record Dates: First submitted 2016-10-29; First posted 2016-11-02 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye; Posterior Blepharitis
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BlephEx treatment (Active Comparator): Treatment with the BlephEx instrument (lid margin exfoliation)
  Interventions: Device: Blephex
- MiBoFlo treatment (Active Comparator): Treatment with the MiboFlo equipment (heat therapy to eyelids)
  Interventions: Device: MiboFlo

INTERVENTIONS:
Device: Blephex — Lid margin exfoliation
  Arms: BlephEx treatment
Device: MiboFlo — Lid warming treatment
  Arms: MiBoFlo treatment

SUMMARY:
The goal of this study is to compare which treatment - BlephEx or MiBoFlo - will be a better option for patients suffering from dry eye secondary to Meibomian Gland dysfunction.

DETAILED DESCRIPTION:
The investigators have previously studied the effect of the BlephEx instrument (debridement of lid debris) in relieving signs and symptoms of blepharitis (Connor CG et al, ARVO 2014). This previous study demonstrated positive results from the BlephEx treatment. Warming the eyelids (e.g., using warm wash cloths) still remains a viable treatment option for this disease. However, patients are often non-compliant with warm compress therapy due to the requirement of performing it at least twice per day. The MiBoflo delivers uniform and consistent amounts of heat to the eyelid. It is suggested that two treatments over 30 days is adequate to relieve signs and symptoms of Meibomian gland dysfunction. This equipment is currently used in optometric practices in this country.

There are no clinical studies comparing BlephEx and MiBoflo as treatment options for blepharitis. Hence, the current study will provide new and useful information on which treatment option may be better for treating blepharitis and Meibomian gland dysfunction. Part of this study will also investigate if a combination of BlephEx and MiBoflo treatments is more beneficial to the patient. The data generated will directly benefit clinical practice and impact several millions of patients who suffer from this Blepharitis and / or Meibomian gland dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Must have dry eye secondary to Meibomian gland dysfunction (posterior blepharitis)

Exclusion Criteria:

* Must not have active ocular surface infections. Must not be currently using steroids or immunosuppression eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Ocular irritation symptoms (OSDI Questionnaire score) | one month

SECONDARY OUTCOMES:
Tear break-up | one month

CONTACTS AND LOCATIONS:
Overall Officials: Srihari Narayanan, OD, PhD, Principal Investigator — University of the Incarnate Word
Locations (1):
- Rosenberg School of Optometry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD to other researchers